CLINICAL TRIAL: NCT06961786
Title: A Phase 1, Open-label, Single-arm Study to Investigate the Safety, Tolerability, and Preliminary Efficacy of TNFa and IL-2 Coding Oncolytic Adenovirus TILT-123 in Combination With Lymphocyte-depleting Chemotherapy and Tumor-infiltrating Lymphocytes in Melanoma Patients.
Brief Title: TNFα and IL-2 Coding Oncolytic Adenovirus TILT-123 With Lymphocyte-depleting Chemotherapy and TILs in the Treatment of Melanoma
Acronym: TUNINTIL-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILT-T216; 2024-514092-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-23; First posted 2025-05-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Melanoma
Keywords: oncolytic virus; TILT; immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILT-123, TILs and chemotherapy (Experimental): TILT-123 in combination with lymphocyte-depleting chemotherapy and TILs
  Interventions: Biological: TILT-123; Biological: TIL; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: TILT-123 — TNFalpha and IL-2 coding oncolytic adenovirus TILT-123
  Other Names: Ad5/3-E2F-d24-hTNFa-IRES-hIL2
Biological: TIL — Adoptive T cell therapy with TILs
  Other Names: Tumor-infiltrating lymphocytes
Drug: Cyclophosphamide — Lymphocyte-depleting chemotherapy
  Other Names: Cytoxan; cyclophosphane
Drug: Fludarabine — Lymphocyte-depleting chemotherapy
  Other Names: Fludara

SUMMARY:
This is an open-label, phase 1 trial evaluating the safety of oncolytic adenovirus TILT-123 in combination with lymphocyte-depleting chemotherapy and TILs in metastatic melanoma patients.

DETAILED DESCRIPTION:
TILT-123 is a tumor-selective replicating oncolytic adenovirus expressing TNFa and IL-2 that is being investigated in several Phase 1 clinical studies in patients with various types of cancer. This is the second study of TILT-123 in patients with metastatic melanoma. Building upon the previous study, TILT-T215, which evaluated the safety and preliminary efficacy of TILT-123 in combination with TILs, Study TILT-T216 will investigate the addition of lymphocyte-depleting chemotherapy to the combination of TILT-123 and TILs. The purpose of lymphodepleting chemotherapy, cyclophosphamide and fludarabine phosphate is to reduce irrelevant T cells and eliminate the regulatory T cells, which are known to be able to inhibit T-cell mediated tumor cell killing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
2. Patients with pathologically confirmed previously treated refractory or recurrent stage 3-4 melanoma, which cannot be treated with curative intent with available therapies.
3. Patients who have had at least 1 prior line of medical treatment (eg, checkpoint inhibitors, kinase inhibitors, IL-2). Multiple prior therapies (eg, surgery, checkpoint inhibitors, kinase inhibitors, IL-2, interferon, chemotherapy, radiation) are allowed.
4. Patients must have a demonstrated WHO/ECOG performance score of 0-1 at screening.
5. A tumor of >9 mm in diameter (typically a minimum of 1 cm3 in volume), without signs of necrosis, must be available for biopsy/operation to enable growing of TILs.
6. At least 1 additional tumor (>14 mm in diameter) must be available for injections and biopsies for correlative analyses. The disease burden must be evaluable according to RECIST 1.1.
7. Patients must have adequate hepatic, cardiac, and renal function as follows:

   1. Platelets ≥ 100,000/µl and < 700,000/µl
   2. Hemoglobin ≥100 g/L
   3. AST and ALT ≤2.5×ULN
   4. GFR >60 mL/min (CKD-EPI)
   5. Leukocytes (WBC) >3.0G/L
   6. Absolute neutrophil count greater than 1500/mm3 without the support of filgrastim
   7. Bilirubin <1.5×ULN
   8. Patients of 60 years or older, or have a history of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, heart block, will undergo cardiac evaluation: LVEF assessment with documented LVEF ≥ 50% by either TTE (trans thoracal echocardiography) or MUGA (multigated acquisition scan). Further cardiac evaluations in patients with cardiac risk factors (e.g. diabetes, hypertension, obesity) will be evaluated by the investigator as deemed necessary.
8. Must be willing to use adequate forms of contraception from screening, during the study, and for a minimum of 90 days after the end of treatment, in accordance with the following:

   1. Woman of childbearing potential: Barrier contraceptive method (ie, condom) must be used in addition to 1 of the following methods: Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections).
   2. Women not of childbearing potential: Barrier contraceptive method (ie, condom) must be used.
   3. Men: Barrier contraceptive method (ie, condom) must be used.
9. Patients must be capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
10. Patients must be capable of understanding and complying with the parameters outlined in the protocol.
11. Patients must have a life expectancy longer than 3 months.
12. Patients must be eligible for adoptive T-cell therapy with Lymphocyte-depleting chemotherapy and TILs.

Exclusion Criteria:

1. History of another active invasive cancer as judged by the investigator within the past 3 years except basal cell carcinoma.
2. Uncontrolled cardiac or vascular diseases.
3. History of heart attack or cerebral stroke within the previous 12 months before screening or is not recovered from a previous heart attack or cerebral stroke.
4. History of hepatic dysfunction, hepatitis, or human immunodeficiency virus.

   1. Patients should be seronegative for HIV antibody.
   2. Patients should be seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
5. History of coagulation disorder.
6. Untreated brain metastases. Treated brain metastases that have not progressed in the 3 months prior to screening are allowed.
7. Concurrent opportunistic and/or active systemic infections.
8. Use of immunosuppressive medications (corticosteroids or drugs used in treatment of autoimmune disease), except for the following, which can be allowed at screening and during the study:

   1. Replacement corticosteroids (eg, if the patient has adrenal insufficiency after prior immunotherapy)
   2. Pulmonary and topical treatments
   3. Prednisone/prednisolone at doses up to 20 mg/day
9. Treated with any anticancer therapy (eg, immunotherapy, signal-transduction inhibitors [eg. BRAF and MEK inhibitors], cytotoxic chemotherapy, radiotherapy, or investigational agents [ie, any drug or therapy that is currently not approved for use in humans]) within 30 days prior to enrollment.
10. Previously treated with any oncolytic adenovirus that was administered IT.
11. Previously treated with adoptive cell therapy.
12. Administered an IMP or device in another clinical study within 30 days prior to baseline.
13. Lactate dehydrogenase value >5×ULN.
14. Allergy to any ingredients present in the IMPs (as listed in the respective IBs).
15. Women of childbearing potential who are pregnant, breastfeeding, or intending to become pregnant.
16. Any other medical condition or laboratory abnormality that, in the judgment of the principal investigator, could increase the risk associated with study participation, interfere with interpretation of study results, or otherwise render study participation inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any (serious and non-serious) Adverse Events | 78 days
  Adverse events
Number of Participants with abnormal laboratory values | 78 days
  Laboratory values
Number of Participants with vital sign abnormalities | 78 days
  Vital signs
Safety assessed by 12- lead electrocardiograms (ECGs) Adverse Events | 78 days
  Clinically significant abnormalities detected in the evaluation (including for example rate, rhythm, axis calculations and interpretation of P, Q, R, S, T U waves, segments and basic ECG calculations) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Principal Investigator — CCIT, Herlev Hospital, Copenhagen University
Locations (1):
- National Center for Cancer Immune Therapy Herlev Hospital, Copenhagen University, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No